CLINICAL TRIAL: NCT04316455
Title: Impact of Self-managed Integrative Yoga Therapy for Older Adults Living With Chronic Pain
Brief Title: Self-managed Integrative Yoga Therapy for Older Adults Living With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarogyam UK (Other)
Collaborators: Hindu Swayamsevak Sangh (UK) (Unknown); Leicester Ageing Together (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AU06
Record Dates: First submitted 2020-03-17; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Integrative Yoga Therapy (Experimental): Participants engaging in a 6-week chronic pain self-management program. Intervention: Integrative Yoga Therapy
  Interventions: Other: Integrative Yoga Therapy

INTERVENTIONS:
Other: Integrative Yoga Therapy — Participants having an hour in-person weekly session with qualified yoga therapist for 6-weeks. At each session, the personalised yoga practices including straightening and relaxing posture of yoga, yoga breathing, Combinations of sound and imagery yoga practices were given and asked to continue practice at home during the week.

SUMMARY:
Chronic pain self-management skills can help patients improve daily functioning and quality of life. The goal of this study is to evaluate chronic pain self-managed Integrative Yoga Therapy intervention delivered in a sample of 25 older adults recruited from community site in Leicester.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent
* Age >= 60 years
* Ambulatory
* Community-living
* Self-reported chronic musculoskeletal pain > 3 months having pain made it difficult to do usual activities
* Ability to attend sessions one in a week for 6-weeks

Exclusion Criteria:

* Serious illness or hospitalisation in last 3-month
* Planned surgery in next six months
* Significant cognitive impairment
* Other severe physical or psychiatric disorder

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-07 (Actual)

PRIMARY OUTCOMES:
Pain severity and interference: Brief Pain Inventory (BPI) questionnaire | From baseline to 6-week post intervention
  Pain severity and interference were evaluated by using the Brief Pain Inventory (BPI) questionnaire.

SECONDARY OUTCOMES:
Participant Global Impression of Change | From baseline to 6-week post intervention
  Participant Global Impression of Change included 2 item the change from baseline
Participant satisfaction: Likert-scale questions | From baseline to 6-week post intervention
  Likert-scale questions score between 1-5 for participant satisfaction with the program (Strongly Agree=1 to Strongly Disagree=5)

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Aarogyam UK; Jaydeep Joshi, BAMS, Study Director — Aarogyam UK; Usha Solanki, Study Chair — Hindu Swayamsevak Sangh (UK); Bharti Mistry, Study Chair — Leicester Ageing Together UK
Locations (1):
- Karyalaya, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided